CLINICAL TRIAL: NCT05968066
Title: Practice of Fluid Therapy in Critically Ill Invasively Ventilated Patients (PRoFLUID)--an International Multicenter Observational Cohort Study
Brief Title: Practice of Fluid Therapy in Critically Ill Invasively Ventilated Patients
Acronym: PRoFLUID
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); Amsterdam UMC, location VUmc (Other); University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: PRoFLUID
Record Dates: First submitted 2023-07-10; First posted 2023-08-01 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Fluid Therapy; Vasopressor Therapy; Critical Illness; Invasive Ventilation
Keywords: Fluid Therapy; Vasopressor; Resuscitation; Deresuscitation; Fluids
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this woldwide observational study is to investigate various aspects of fluid and vasopressor therapy in critically ill invasively ventilated patients. The main questions it aims to answer are:

* What is the global current practice of fluid and vasopressor therapy?
* What are associations between this practice and clinical outcomes?

Participating intensive care units will gather detailed information about fluid and vasopressor therapy prescribed to participants. Participating intensive care units will also gather information about participant outcomes such as duration of invasive ventilation, length of stay and mortality

DETAILED DESCRIPTION:
Rationale:

The worldwide practice of fluid and vasopressor therapy in critically ill invasively ventilated patients is uncertain. Indeed, it is unclear whether there is a difference in fluid and vasopressor therapy in these patients between Low- and Middle-income Countries (LMICs) and High-income Countries (HICs).

Objective:

To determine various aspects of fluid and vasopressor therapy in critically ill invasively ventilated patients in LMICs and HICs.

Hypothesis:

There is substantial worldwide variation in practice of fluid and vasopressor therapy in critically ill invasively ventilated patients.

Study design:

International, multicenter, observational study in critically ill invasively ventilated patients; data are captured during a predefined period per geographic region or country.

Study population:

Critically ill invasively ventilated patients.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Because of the observational design of the study using routinely collected data, there is no additional burden for the patient. Collection of data from ICU charts or electronic medical records systems is of no risk to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a participating intensive care unit;
* Receiving invasive ventilation; and
* Duration of ventilation > 24 hours.

Exclusion Criteria:

* Age < 16 years;
* Patients transferred under invasive ventilation from another intensive care unit.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill invasively ventilated patients that receive ventilation for at least 24 hours.
Sampling Method: Probability Sample
Enrollment: 2508 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Composite of various aspects of fluid therapy | seven days
  Including total volumes of types of fluids administered in the first three days after ICU admission and total volume of fluids infused in the first seven days of ICU admission

SECONDARY OUTCOMES:
Timing of start of continuous administration of vasopressors. | seven days
  Timing of start of vasopressors from ICU admission in minutes per administration route (i.e. central versus peripheral)
Duration of vasopressor therapy | seven days
  In days
Types of vasopressors | seven days
  The type (i.e. noradrenaline, vasopressin, adrenaline) of vasopressors that are prescribed
Concentration of types of vasopressors | seven days
  The concentration (i.e. in µg/ml) of vasopressors that are prescribed per administration route
Timing of start of administered diuretics. | seven days
  Time between start of invasive ventilation and administration of diuretics in days
Duration of diuretic therapy | seven days
  In days
Types of diuretics | seven days
  The type of diuretics that are prescribed
Bolus or continous infusion of diuretics | seven days
Cumulative fluid balances | seven days
Daily urine output | seven days
Incidence of atrial arrythmias | 7 days
Incidence of acute respiratory distress syndrome | 7 days
Incidence of renal replacement therapy | 7 days
Incidence of need for renal replacement therapy at ICU discharge. | 90 days
Typical ICU outcomes; e.g. duration of ventilation, lengths of stay in ICU and hospital and, mortality in the ICU and hospital | 90 days

OTHER OUTCOMES:
Pre-defined subgroup analysis in patients admitted with burns | 90 days
  All aforementioned outcomes in patients with burns
Pre-defined subgroup analysis in patients admitted with acute respiratory distress syndrome | 90 days
  All aforementioned outcomes in patients with acute respiratory distress syndrome
Pre-defined subgroup analysis in patients admitted with sepsis | 90 days
  All aforementioned outcomes in patients with sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Pieter R. Tuinman, MD, Principal Investigator — Amsterdam UMC, location VUmc; Frederique Paulus, Professor, Principal Investigator — Amsterdam UMC, location AMC; Marcus J. Schultz, Professor, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] PRoFLUID-Investigators. Practice of Fluid and Vasopressor Therapy in Critically Ill Invasively Ventilated Patients (PRoFLUID)-study protocol for an international multicenter observational cohort study. Ann Transl Med. 2024 Oct 20;12(5):92. doi: 10.21037/atm-23-1957. Epub 2024 Sep 12. PMID 39507456

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-09-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT05968066/SAP_000.pdf